CLINICAL TRIAL: NCT01049035
Title: Safety and Immunogenicity of a Quadrivalent Meningococcal Conjugate Vaccine Administered in Infants and Toddlers
Brief Title: A Study of a Quadrivalent Meningococcal Tetanus Protein Conjugate Vaccine in Infants and Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET39; UTN: U1111-1112-2593 (Other: WHO)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal Infection; Neisseria meningitidis; Tetravalent Meningococcal Vaccine
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Tetanus Toxoid; Vaccines, Combined; pentacel; Rubella Vaccine; Herpes Zoster Vaccine; Chickenpox Vaccine; Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine; 13-valent pneumococcal vaccine; CRM197 (non-toxic variant of diphtheria toxin); Rotavirus Vaccines; RotaTeq; RIX4414 vaccine; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months (Experimental): Participants aged 2 months (at the time of enrollment) received Quadrivalent Meningococcal Polysaccharide (A, C, Y, and W-135) Tetanus Protein (MenACYW) Conjugate vaccine at the age of Months 2, 4, 6, and a booster vaccination at the age of Month 12 along with Prevnar 7 or Prevnar 13 vaccine at the age of Months 2, 4, 6, and 12, Pentacel and Rotavirus vaccines at the age of Months 2, 4, and 6, Hepatitis-B vaccine at the age of Months 2 and 6, and M-M-RII and VARIVAX vaccines at the age of 12 months.
  Interventions: Biological: Quadrivalent Meningococcal Polysaccharide (A, C, Y, and W-135) Tetanus Protein Conjugate; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined); Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live; Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine
- Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months (Experimental): Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of Months 2, 4, 6, and a booster vaccination at the age of Month 15 along with Prevnar 7 or 13 vaccine at the age of Months 2, 4, 6, and 12, Rotavirus vaccine at the age of Months 2, 4, and 6, Hepatitis-B vaccine at the age of Months 2 and 6, M-M-RII and VARIVAX vaccines at the age of Month 12, and Pentacel vaccine at the age of Months 2, 4, 6, and 15.
  Interventions: Biological: Quadrivalent Meningococcal Polysaccharide (A, C, Y, and W-135) Tetanus Protein Conjugate; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined); Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live; Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine
- Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months (Experimental): Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of Months 2, 4 and a booster vaccination at the age of Month 12 along with Pentacel and Rotavirus vaccines at the age of Months 2, 4, and 6, Hepatitis-B vaccine at the age of Months 2 and 6, M-M-RII and VARIVAX vaccines at the age of Month 12, and Prevnar 7 or 13 vaccine at the age of Months 2, 4, 6, and 12.
  Interventions: Biological: Quadrivalent Meningococcal Polysaccharide (A, C, Y, and W-135) Tetanus Protein Conjugate; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined); Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live; Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine
- Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months (Experimental): Participants aged 6 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of Month 6 along with Pentacel, Prevnar 7 or 13, Hepatitis-B and Rotavirus vaccines, and a booster vaccination of MenACYW at the age of Month 12 along with M-M-RII and VARIVAX vaccines. Before enrollment, participants were vaccinated with Pentacel, Prevnar, and Rotavirus vaccines at the age of Months 2 and 4, and Hepatitis-B vaccine at the age of Month 2.
  Interventions: Biological: Quadrivalent Meningococcal Polysaccharide (A, C, Y, and W-135) Tetanus Protein Conjugate; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined); Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live; Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine
- Group 5: MenACYW Conjugate Vaccine: Month 12 (Experimental): Participants aged 12 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of 12 months along with Prevnar 7 or 13, M-M-RII, and VARIVAX vaccines. Before enrollment, participants were vaccinated with Pentacel, Prevnar, and Rotavirus vaccines at the age of Months 2, 4, and 6, and Hepatitis-B vaccine at the age of Months 2 and 6.
  Interventions: Biological: Quadrivalent Meningococcal Polysaccharide (A, C, Y, and W-135) Tetanus Protein Conjugate; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined); Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live; Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine
- Group 6: Control: 2, 4, 6, and 12 Months (Other): Participants aged 2 months (at the time of enrollment) received Pentacel and Rotavirus vaccines at the age of Months 2, 4, and 6, Hepatitis-B vaccine at the age of Months 2 and 6, Prevnar 7 or 13 vaccine at the age of Months 2, 4, 6, and 12 and M-M-RII and VARIVAX vaccines at the age of 12 months.
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined); Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live; Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine
- Group 7: Control: 2, 4, 6, 12, and 15 Months (Other): Participants aged 2 months (at the time of enrollment) received Rotavirus vaccine at the age of Months 2, 4, and 6, Hepatitis-B vaccine at the age of Months 2 and 6, Prevnar 7 or 13 vaccine at the age of Months 2, 4, 6, and 12, and M-M-RII and VARIVAX vaccines at the age of 12 months, and Pentacel vaccine at the age of Months 2, 4, 6, and 15.
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined); Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live; Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein); Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine

INTERVENTIONS:
Biological: Quadrivalent Meningococcal Polysaccharide (A, C, Y, and W-135) Tetanus Protein Conjugate — 0.5 milliliter (mL), Intramuscular (IM) injection
  Other Names: TetraMen-T
  Arms: Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months; Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months; Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months; Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months; Group 5: MenACYW Conjugate Vaccine: Month 12
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus B Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined) — 0.5 mL, IM injection
  Other Names: Pentacel
Biological: M-M-RII-Measles, Mumps, and Rubella Virus Vaccine Live — 0.5 mL, Subcutaneous (SC) injection
Biological: Varicella Virus Vaccine Live — 0.5 mL, SC injection
  Other Names: Varivax
Biological: Pneumococcal 7-valent Conjugate Vaccine (Diphtheria CRM197 Protein) — 0.5 mL, IM injection
  Other Names: Prevnar
Biological: Pneumococcal 13-valent Conjugate Vaccine (Diphtheria CRM197 Protein) — 0.5 mL, IM injection
  Other Names: Prevnar 13
Biological: Rotavirus Vaccine — oral
  Other Names: RotaTeq/ROTARIX
Biological: Hepatitis B Vaccine — 0.5 mL, IM injection
  Other Names: Engerix-B/Recombivax-HB

SUMMARY:
The purpose of this study was to evaluate the optimal vaccination schedule for a Quadrivalent Meningococcal Polysaccharide (A, C, Y and W-135) Tetanus Protein Conjugate Vaccine (MenACYW Conjugate vaccine) in order to provide an effective protein conjugate quadrivalent meningococcal vaccine in the population with the highest incidence of disease.

Objectives:

* To describe the safety profile of MenACYW Conjugate vaccine administered at 5 different schedules and concomitantly with routine pediatric vaccinations.
* To describe the immunogenicity profile of MenACYW Conjugate vaccine administered at 5 different schedules and concomitantly with routine pediatric vaccinations.
* To describe the immunogenicity profiles of selected licensed pediatric vaccines (Pentacel, Prevnar, M-M-RII, and Varivax) when administered either concomitantly with or without MenACYW Conjugate vaccine.

DETAILED DESCRIPTION:
Participants received study vaccinations beginning at age 2, 6, 12, or 15 months, depending on the assigned schedule in their randomized groups. All participants underwent safety and immunogenicity assessments according to the schedule for their assigned group.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1, 2, 3, 6, and 7: Aged 42 to 89 days on the day of inclusion; Group 4: Aged 6 months (180 days ± 14 days) on the day of inclusion; Group 5: Aged 12 months (365 days + 14 days) on the day of inclusion.
* Born at full term of pregnancy (greater than or equal to [≥] 37 weeks) and with a birth weight ≥2.5 kilogram (kg).
* Informed consent form had been signed and dated by the parent or other legally acceptable representative.
* Participant and parent/guardian were able to attend all scheduled visits and to be complied with all trial procedures.
* Group 4 only: Prior receipt of Pentacel and Prevnar at 2 and 4 months; 1 or 2 doses of rotavirus vaccine; and 2 or 3 previous doses of hepatitis B vaccine.

Group 5 only: Prior receipt of Pentacel and Prevnar at 2, 4, and 6 months; 2 or 3 doses of rotavirus vaccine; and 3 previous doses of hepatitis B vaccine.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination, with the exception of influenza vaccine, which may be received 14 days before or after MenACYW Conjugate vaccine.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine.
* Receipt of blood or blood-derived products in the past 30 days, which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks).
* Known personal or maternal seropositivity for human immunodeficiency virus (HIV), hepatitis B vaccine, or hepatitis C, as reported by the parent/guardian.
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia, as reported by the parent/guardian.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* History of seizures.
* Personal or family history of Guillain-Barré Syndrome (GBS).
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.

Temporary contraindications were resolved before vaccination:

* Febrile illness (temperature ≥38.0 degree Celsius [≥100.4 degree Fahrenheit]) or moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination.
* Group 5 only: Receipt of oral or injected antibiotic therapy within the 72 hours prior to the study blood draw. Topical antibiotics or antibiotic drops were not included in this exclusion criterion. (Note: This did not applied to the other groups at this time, as they did not have a blood draw within 30 days of the initial visit.).

Ages: 42 Days to 365 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 580 (Actual)
Dates: Start 2009-12-16 (Actual); Primary Completion 2012-02-13 (Actual); Study Completion 2012-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (23):
- United States (23):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Huntington Beach, California
  - Marietta, Georgia
  - Woodstock, Georgia
  - Bardstown, Kentucky
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Bossier City, Louisiana
  - Clyde, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Barnwell, South Carolina
  - Clarksville, Tennessee
  - Fort Worth, Texas
  - Layton, Utah
  - Orem, Utah
  - Springville, Utah
  - Midlothian, Virginia
  - Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Cornish MJ, Hedrick JA, Gabrielsen AA, Johnson AD, Miriam Pina L, Rehm C, Pan J, Neveu D, Da Costa X, Jordanov E, Dhingra MS. Safety and immunogenicity of an investigational quadrivalent meningococcal tetanus toxoid conjugate vaccine (MenACYW-TT) co-administered with routine pediatric vaccines in infants and toddlers: A Phase II study. Vaccine. 2022 Mar 1;40(10):1421-1438. doi: 10.1016/j.vaccine.2022.01.050. Epub 2022 Feb 7. PMID 35144847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from 16 December 2009 to 13 February 2012 at 21 active sites in the United States.
Pre-assignment Details: A total of 580 participants who met all inclusion and none of the exclusion criteria were enrolled and randomized in the study.
Groups:
- Group 5: MenACYW Conjugate Vaccine: 12 Months: Participants aged 12 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of 12 months along with Prevnar 7 or 13, M-M-RII, and VARIVAX vaccines. Before enrollment, participants were vaccinated with Pentacel, Prevnar, and Rotavirus vaccines at the age of Months 2, 4, and 6, and Hepatitis-B vaccine at the age of Months 2 and 6.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 5: MenACYW Conjugate Vaccine: 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Started | 107 | 108 | 107 | 75 | 75 | 54 | 54
Safety Population (Participants who received at least 1 dose of study/control vaccine and had safety data available.) | 104 | 102 | 100 | 74 | 70 | 52 | 49
Completed | 74 | 87 | 80 | 64 | 71 | 42 | 39
Not Completed | 33 | 21 | 27 | 11 | 4 | 12 | 15
Not completed — Serious adverse event | 0 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Other adverse event (AE) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance with the protocol | 12 | 6 | 14 | 5 | 3 | 4 | 10
Not completed — Lost to Follow-up | 5 | 4 | 4 | 1 | 0 | 3 | 3
Not completed — Voluntary withdrawal not due to an AE | 16 | 10 | 8 | 2 | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months: Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of Months 2, 4, 6, and a booster vaccination at the age of Month 12 along with Prevnar 7 or Prevnar 13 vaccine at the age of Months 2, 4, 6, and 12, Pentacel and Rotavirus vaccines at the age of Months 2, 4, and 6, Hepatitis-B vaccine at the age of Months 2 and 6, and M-M-RII and VARIVAX vaccines at the age of 12 months.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 5: MenACYW Conjugate Vaccine: 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months | Total
Number analyzed (Participants) | 107 | 108 | 107 | 75 | 75 | 54 | 54 | 580
Age, Continuous [Mean (Standard Deviation); unit: months] | 2.19 (0.261) | 2.20 (0.259) | 2.23 (0.296) | 6.23 (0.148) | 12.4 (0.136) | 2.18 (0.217) | 2.20 (0.268) | 4.04 (3.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 47 | 38 | 31 | 24 | 20 | 277
  Male | 50 | 48 | 60 | 37 | 44 | 30 | 34 | 303
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Black | 10 | 11 | 15 | 9 | 4 | 4 | 10 | 63
  Caucasian | 86 | 73 | 78 | 60 | 60 | 42 | 33 | 432
  Hispanic | 4 | 4 | 7 | 0 | 3 | 2 | 2 | 22
  American Indian or Alaska Native | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 4
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Other | 7 | 17 | 5 | 5 | 7 | 6 | 8 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Serum Bactericidal Assay (SBA) Using Human Complement (SBA-HC) Titer Greater or Than Equal to (≥) 1:8 and ≥1:4: Groups 1, 2, 3, 4, 6, and 7 - Primary Series Per-protocol Population (PPP)
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. The PPP consisted of all participants included in the trial who received at least one dose of study or control vaccine, excluding those who did not meet all protocol-specified inclusion/exclusion criteria, did not receive the correct number of doses of the investigational vaccine, received a vaccine other than the one that he/she was randomized to receive, did not provide a post-dose serology sample in the proper time window, received a protocol-restricted therapy, medication or vaccine, was on systemic antibiotics within 3 days prior to study blood draw, had no serology sample or did not produce at least one valid test result, did not receive vaccine in the proper time window. Primary series PPP was defined as the PPP which was used for reporting data of time points prior to 12 months of age.
Time Frame: Groups 1, 2, 4, 6, and 7: at the age of 7 months; Group 3: at the age of 5 months
Population: Primary series PPP. 'Number analyzed'=number of participants with available data for specified categories and '0' in number analyzed field signifies none of the participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 78 | 81 | 77 | 61 | 45 | 35
percentage of participants
  Serogroup A- at 5 months of age: ≥1:4: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup A- at 5 months of age: ≥1:4 |  |  | 83.1 [72.9 to 90.7] |  |  |
  Serogroup A- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup A- at 5 months of age: ≥1:8 |  |  | 74.0 [62.8 to 83.4] |  |  |
  Serogroup A- at 7 months of age: ≥1:4: number analyzed (Participants) | 77 | 81 | 0 | 58 | 44 | 35
  Serogroup A- at 7 months of age: ≥1:4 | 80.5 [69.9 to 88.7] | 80.2 [69.9 to 88.3] |  | 75.9 [62.8 to 86.1] | 15.9 [6.6 to 30.1] | 25.7 [12.5 to 43.3]
  Serogroup A- at 7 months of age: ≥1:8: number analyzed (Participants) | 77 | 81 | 0 | 58 | 44 | 35
  Serogroup A- at 7 months of age: ≥1:8 | 71.4 [60.0 to 81.2] | 66.7 [55.3 to 76.8] |  | 62.1 [48.4 to 74.5] | 4.5 [0.6 to 15.5] | 2.9 [0.1 to 14.9]
  Serogroup C- at 5 months of age: ≥1:4: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup C- at 5 months of age: ≥1:4 |  |  | 97.4 [90.9 to 99.7] |  |  |
  Serogroup C- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup C- at 5 months of age: ≥1:8 |  |  | 94.8 [87.2 to 98.6] |  |  |
  Serogroup C- at 7 months of age: ≥1:4: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup C- at 7 months of age: ≥1:4 | 96.2 [89.2 to 99.2] | 93.8 [86.2 to 98.0] |  | 90.2 [79.8 to 96.3] | 11.1 [3.7 to 24.1] | 17.1 [6.6 to 33.6]
  Serogroup C- at 7 months of age: ≥1:8: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup C- at 7 months of age: ≥1:8 | 92.3 [84.0 to 97.1] | 92.6 [84.6 to 97.2] |  | 88.5 [77.8 to 95.3] | 2.2 [0.1 to 11.8] | 2.9 [0.1 to 14.9]
  Serogroup Y- at 5 months of age: ≥1:4: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup Y- at 5 months of age: ≥1:4 |  |  | 83.1 [72.9 to 90.7] |  |  |
  Serogroup Y- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup Y- at 5 months of age: ≥1:8 |  |  | 75.3 [64.2 to 84.4] |  |  |
  Serogroup Y- at 7 months of age: ≥1:4: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup Y- at 7 months of age: ≥1:4 | 97.4 [91.0 to 99.7] | 93.8 [86.2 to 98.0] |  | 29.5 [18.5 to 42.6] | 8.9 [2.5 to 21.2] | 11.4 [3.2 to 26.7]
  Serogroup Y- at 7 months of age: ≥1:8: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup Y- at 7 months of age: ≥1:8 | 89.7 [80.8 to 95.5] | 91.4 [83.0 to 96.5] |  | 24.6 [14.5 to 37.3] | 6.7 [1.4 to 18.3] | 5.7 [0.7 to 19.2]
  Serogroup W-135- at 5 months of age: ≥1:4: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup W-135- at 5 months of age: ≥1:4 |  |  | 92.2 [83.8 to 97.1] |  |  |
  Serogroup W-135- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup W-135- at 5 months of age: ≥1:8 |  |  | 84.4 [74.4 to 91.7] |  |  |
  Serogroup W-135- at 7 months of age: ≥1:4: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup W-135- at 7 months of age: ≥1:4 | 98.7 [93.1 to 100.0] | 98.8 [93.3 to 100.0] |  | 42.6 [30.0 to 55.9] | 11.1 [3.7 to 24.1] | 11.4 [3.2 to 26.7]
  Serogroup W-135- at 7 months of age: ≥1:8: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup W-135- at 7 months of age: ≥1:8 | 94.9 [87.4 to 98.6] | 96.3 [89.6 to 99.2] |  | 24.6 [14.5 to 37.3] | 2.2 [0.1 to 11.8] | 2.9 [0.1 to 14.9]

2. Primary Outcome: Percentage of Participants With an Serum Bactericidal Assay Using Human Complement Titer ≥1:8 and ≥1:4: Groups 1, 2, 3, 4, 6, and 7 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. PPP consisted of all participants included in the trial who received at least one dose of study or control vaccine, excluding those who did not meet all protocol-specified inclusion/exclusion criteria, did not received the correct number of doses of the investigational vaccine, received a vaccine other than the one that he/she was randomized to receive, did not provided a post-dose serology sample in the proper time window, received a protocol-restricted therapy, medication or vaccine, was on systemic antibiotics within 3 days prior to study blood draw, had no serology sample or did not produce at least one valid test result, did not receive vaccine in the proper time window. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: Groups 1, 3, 4, and 6: at the age of 13 months; Groups 2 and 7: at the age of 16 months
Population: Booster PPP. Here, 'Number analyzed'=number of participants with available data for specified categories and '0' in number analyzed field signifies none of the participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49 | 27 | 28
percentage of participants
  Serogroup A- at 13 months of age: ≥1:4: number analyzed (Participants) | 59 | 0 | 55 | 46 | 25 | 0
  Serogroup A- at 13 months of age: ≥1:4 | 94.9 [85.9 to 98.9] |  | 96.4 [87.5 to 99.6] | 100.0 [92.3 to 100.0] | 28.0 [12.1 to 49.4] |
  Serogroup A- at 13 months of age: ≥1:8: number analyzed (Participants) | 59 | 0 | 55 | 46 | 25 | 0
  Serogroup A- at 13 months of age: ≥1:8 | 94.9 [85.9 to 98.9] |  | 94.5 [84.9 to 98.9] | 100.0 [92.3 to 100.0] | 12.0 [2.5 to 31.2] |
  Serogroup A- at 16 months of age: ≥1:4: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup A- at 16 months of age: ≥1:4 |  | 96.9 [89.2 to 99.6] |  |  |  | 30.8 [14.3 to 51.8]
  Serogroup A- at 16 months of age: ≥1:8: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup A- at 16 months of age: ≥1:8 |  | 93.8 [84.8 to 98.3] |  |  |  | 15.4 [4.4 to 34.9]
  Serogroup C- at 13 months of age: ≥1:4: number analyzed (Participants) | 59 | 0 | 55 | 46 | 26 | 0
  Serogroup C- at 13 months of age: ≥1:4 | 94.9 [85.9 to 98.9] |  | 94.5 [84.9 to 98.9] | 100.0 [92.3 to 100.0] | 30.8 [14.3 to 51.8] |
  Serogroup C- at 13 months of age: ≥1:8: number analyzed (Participants) | 59 | 0 | 55 | 46 | 26 | 0
  Serogroup C- at 13 months of age: ≥1:8 | 94.9 [85.9 to 98.9] |  | 90.9 [80.0 to 97.0] | 100.0 [92.3 to 100.0] | 7.7 [0.9 to 25.1] |
  Serogroup C- at 16 months of age: ≥1:4: number analyzed (Participants) | 0 | 65 | 0 | 0 | 0 | 26
  Serogroup C- at 16 months of age: ≥1:4 |  | 98.5 [91.7 to 100.0] |  |  |  | 34.6 [17.2 to 55.7]
  Serogroup C- at 16 months of age: ≥1:8: number analyzed (Participants) | 0 | 65 | 0 | 0 | 0 | 26
  Serogroup C- at 16 months of age: ≥1:8 |  | 96.9 [89.3 to 99.6] |  |  |  | 3.8 [0.1 to 19.6]
  Serogroup Y- at 13 months of age: ≥1:4: number analyzed (Participants) | 59 | 0 | 54 | 46 | 26 | 0
  Serogroup Y- at 13 months of age: ≥1:4 | 100.0 [93.9 to 100.0] |  | 100.0 [93.4 to 100.0] | 100.0 [92.3 to 100.0] | 11.5 [2.4 to 30.2] |
  Serogroup Y- at 13 months of age: ≥1:8: number analyzed (Participants) | 59 | 0 | 54 | 46 | 26 | 0
  Serogroup Y- at 13 months of age: ≥1:8 | 100.0 [93.9 to 100.0] |  | 98.1 [90.1 to 100.0] | 97.8 [88.5 to 99.9] | 3.8 [0.1 to 19.6] |
  Serogroup Y- at 16 months of age: ≥1:4: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup Y- at 16 months of age: ≥1:4 |  | 100.0 [94.4 to 100.0] |  |  |  | 11.5 [2.4 to 30.2]
  Serogroup Y- at 16 months of age: ≥1:8: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup Y- at 16 months of age: ≥1:8 |  | 100.0 [94.4 to 100.0] |  |  |  | 3.8 [0.1 to 19.6]
  Serogroup W-135- at 13 months of age: ≥1:4: number analyzed (Participants) | 59 | 0 | 54 | 46 | 25 | 0
  Serogroup W-135- at 13 months of age: ≥1:4 | 100.0 [93.9 to 100.0] |  | 100.0 [93.4 to 100.0] | 100.0 [92.3 to 100.0] | 8.0 [1.0 to 26.0] |
  Serogroup W-135- at 13 months of age: ≥1:8: number analyzed (Participants) | 59 | 0 | 54 | 46 | 25 | 0
  Serogroup W-135- at 13 months of age: ≥1:8 | 100.0 [93.9 to 100.0] |  | 98.1 [90.1 to 100.0] | 97.8 [88.5 to 99.9] | 4.0 [0.1 to 20.4] |
  Serogroup W-135- at 16 months of age: ≥1:4: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup W-135- at 16 months of age: ≥1:4 |  | 100.0 [94.4 to 100.0] |  |  |  | 3.8 [0.1 to 19.6]
  Serogroup W-135- at 16 months of age: ≥1:8: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup W-135- at 16 months of age: ≥1:8 |  | 100.0 [94.4 to 100.0] |  |  |  | 3.8 [0.1 to 19.6]

3. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement Titer ≥1:8 and ≥1:4: Group 5 - Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. PPP consisted of all participants included in the trial who received at least one dose of study or control vaccine, excluding those who did not meet all protocol-specified inclusion/exclusion criteria, did not received the correct number of doses of the investigational vaccine, received a vaccine other than the one that he/she was randomized to receive, did not provided a post-dose serology sample in the proper time window, received a protocol-restricted therapy, medication or vaccine, was on systemic antibiotics within 3 days prior to study blood draw, had no serology sample or did not produce at least one valid test result, did not receive vaccine in the proper time window.
Time Frame: At the age of 13 months
Population: Analysis was performed on PPP. Here, 'Number analyzed'=participants with available data for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 62
percentage of participants
  Serogroup A: ≥1:4: number analyzed (Participants) | 59
  Serogroup A: ≥1:4 | 81.4 [69.1 to 90.3]
  Serogroup A: ≥1:8: number analyzed (Participants) | 59
  Serogroup A: ≥1:8 | 74.6 [61.6 to 85.0]
  Serogroup C: ≥1:4: number analyzed (Participants) | 61
  Serogroup C: ≥1:4 | 96.7 [88.7 to 99.6]
  Serogroup C: ≥1:8: number analyzed (Participants) | 61
  Serogroup C: ≥1:8 | 90.2 [79.8 to 96.3]
  Serogroup Y: ≥1:4: number analyzed (Participants) | 61
  Serogroup Y: ≥1:4 | 60.7 [47.3 to 72.9]
  Serogroup Y: ≥1:8: number analyzed (Participants) | 61
  Serogroup Y: ≥1:8 | 47.5 [34.6 to 60.7]
  Serogroup W-135: ≥1:4: number analyzed (Participants) | 59
  Serogroup W-135: ≥1:4 | 69.5 [56.1 to 80.8]
  Serogroup W-135: ≥1:8: number analyzed (Participants) | 59
  Serogroup W-135: ≥1:8 | 54.2 [40.8 to 67.3]

4. Primary Outcome: Percentage of Participants With SBA-HC Pre-booster Titer ≥1:8 Who Then Achieved ≥4-Fold Rise in SBA-HC Titer After Booster Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. Pre-booster titer was defined as titer values reported before the age of 12 months. Percentage of participants whose pre-booster titer was ≥1:8 and achieved ≥4-fold rise in each meningococcal serogroups antibody titer (30-days post booster vaccination) were reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: Groups 1, 3, and 4: 30 days post-vaccination at the age of 12 months (i.e. at the age of 13 months); Group 2: 30 days post-vaccination at the age of 15 months (i.e. at the age of 16 months)
Population: Analysis was performed on booster PPP. Here, 'Number analyzed'=participants with available data for specified category. Data for this outcome measure were not planned to be collected and analyzed for Groups 6 and 7, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
percentage of participants
  Serogroup A: number analyzed (Participants) | 23 | 20 | 15 | 11
  Serogroup A | 82.6 [61.2 to 95.0] | 85.0 [62.1 to 96.8] | 66.7 [38.4 to 88.2] | 100.0 [71.5 to 100.0]
  Serogroup C: number analyzed (Participants) | 33 | 35 | 26 | 39
  Serogroup C | 97.0 [84.2 to 99.9] | 97.1 [85.1 to 99.9] | 92.3 [74.9 to 99.1] | 100.0 [91.0 to 100.0]
  Serogroup Y: number analyzed (Participants) | 49 | 59 | 42 | 39
  Serogroup Y | 83.7 [70.3 to 92.7] | 91.5 [81.3 to 97.2] | 81.0 [65.9 to 91.4] | 94.9 [82.7 to 99.4]
  Serogroup W-135: number analyzed (Participants) | 52 | 58 | 43 | 42
  Serogroup W-135 | 94.2 [84.1 to 98.8] | 84.5 [72.6 to 92.7] | 90.7 [77.9 to 97.4] | 88.1 [74.4 to 96.0]

5. Primary Outcome: Percentage of Participants With SBA-HC Pre-vaccination Titer ≥1:8 Who Then Achieved ≥4-fold Rise in SBA-HC Titer After Vaccination: Group 5 - Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. Pre-vaccination titer was defined as titer values reported before the age of 12 months. Percentage of participants whose pre-vaccination titer was ≥1:8 and achieved ≥4-fold rise in each meningococcal serogroups antibody titer (30 days post-vaccination) were reported.
Time Frame: 30 days post-vaccination at the age of 12 months (i.e. at the age of 13 months)
Population: Analysis was performed on PPP. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure and '0' in the number analyzed field signifies none of the participants had pre-vaccination titer ≥1:8.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 3
percentage of participants
  Serogroup A | 33.3 [0.8 to 90.6]
  Serogroup C | 66.7 [9.4 to 99.2]
  Serogroup Y: number analyzed (Participants) | 0
  Serogroup W-135: number analyzed (Participants) | 0

6. Primary Outcome: Percentage of Participants With SBA-HC Pre-booster Titer Less Than (<) 1:8 Who Then Achieved ≥4-Fold Rise in SBA-HC After Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. Pre-booster titer was defined as titer values reported before the age of 12 months. Percentage of participants whose pre-booster titer was <1:8 and achieved ≥4-fold rise in each meningococcal serogroups antibody titer (30-days post booster vaccination) were reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: as for outcome 4
Population: Analysis was performed on booster PPP. Here, 'Number analyzed'=participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Groups 6 and 7, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
percentage of participants
  Serogroup A: number analyzed (Participants) | 33 | 42 | 38 | 33
  Serogroup A | 84.8 [68.1 to 94.9] | 85.7 [71.5 to 94.6] | 92.1 [78.6 to 98.3] | 97.0 [84.2 to 99.9]
  Serogroup C: number analyzed (Participants) | 24 | 29 | 27 | 6
  Serogroup C | 87.5 [67.6 to 97.3] | 93.1 [77.2 to 99.2] | 74.1 [53.7 to 88.9] | 83.3 [35.9 to 99.6]
  Serogroup Y: number analyzed (Participants) | 8 | 4 | 10 | 6
  Serogroup Y | 87.5 [47.3 to 99.7] | 100.0 [39.8 to 100.0] | 90.0 [55.5 to 99.7] | 83.3 [35.9 to 99.6]
  Serogroup W-135: number analyzed (Participants) | 5 | 5 | 9 | 3
  Serogroup W-135 | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 88.9 [51.8 to 99.7] | 66.7 [9.4 to 99.2]

7. Primary Outcome: Percentage of Participants With SBA-HC Pre-Vaccination Titer <1:8 Who Then Achieved ≥4-Fold Rise in SBA-HC Titer After Vaccination: Group 5 - Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. Percentage of participants with pre-vaccination titer <1:8 and achieved ≥4-fold rise in each meningococcal serogroups antibody titer (30-days post vaccination) were reported.
Time Frame: 30 days post-vaccination at the age of 12 months (i.e. at the age of 13 months)
Population: Analysis was performed on PPP. Here, 'Number analyzed'=participants with available data for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 62
percentage of participants
  Serogroup A: number analyzed (Participants) | 55
  Serogroup A | 60.0 [45.9 to 73.0]
  Serogroup C: number analyzed (Participants) | 57
  Serogroup C | 87.7 [76.3 to 94.9]
  Serogroup Y: number analyzed (Participants) | 60
  Serogroup Y | 35.0 [23.1 to 48.4]
  Serogroup W-135: number analyzed (Participants) | 58
  Serogroup W-135 | 29.3 [18.1 to 42.7]

8. Primary Outcome: Serum Bactericidal Assay Using Human Complement Geometric Mean Titers (GMTs): Groups 1, 2, 3, 4, 6, and 7 - Primary Series Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. Primary series PPP was defined as the PPP which was used for reporting data of time points prior to 12 months of age.
Time Frame: Groups 1, 2, 4, 6, and 7: at the age of 7 months, Group 3: at the age of 5 months
Population: Primary series PPP. Here, 'Number analyzed'=participants with available data for specified categories and '0' in number analyzed field signifies none of the participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 78 | 81 | 77 | 61 | 45 | 35
titers (1/dilution)
  Serogroup A- at 5 months of age: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup A- at 5 months of age |  |  | 16.3 [11.9 to 22.2] |  |  |
  Serogroup A- at 7 months of age: number analyzed (Participants) | 77 | 81 | 0 | 58 | 44 | 35
  Serogroup A- at 7 months of age | 14.8 [10.7 to 20.4] | 16.1 [11.3 to 23.1] |  | 9.8 [6.9 to 13.8] | 2.4 [2.0 to 2.9] | 2.5 [2.1 to 3.0]
  Serogroup C- at 5 months of age: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup C- at 5 months of age |  |  | 103.1 [72.7 to 146.4] |  |  |
  Serogroup C- at 7 months of age: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup C- at 7 months of age | 101.6 [69.9 to 147.7] | 93.3 [63.9 to 136.2] |  | 40.2 [27.1 to 59.6] | 2.3 [1.9 to 2.8] | 2.3 [2.0 to 2.7]
  Serogroup Y- at 5 months of age: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup Y- at 5 months of age |  |  | 17.8 [12.8 to 24.7] |  |  |
  Serogroup Y- at 7 months of age: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup Y- at 7 months of age | 33.8 [25.6 to 44.5] | 39.3 [29.5 to 52.4] |  | 3.3 [2.6 to 4.0] | 2.4 [1.9 to 3.0] | 2.3 [2.0 to 2.8]
  Serogroup W-135- at 5 months of age: number analyzed (Participants) | 0 | 0 | 77 | 0 | 0 | 0
  Serogroup W-135- at 5 months of age |  |  | 23.4 [17.2 to 31.7] |  |  |
  Serogroup W-135- at 7 months of age: number analyzed (Participants) | 78 | 81 | 0 | 61 | 45 | 35
  Serogroup W-135- at 7 months of age | 50.8 [39.4 to 65.6] | 47.4 [36.6 to 61.5] |  | 3.7 [2.9 to 4.7] | 2.4 [1.9 to 3.0] | 2.2 [2.0 to 2.4]

9. Primary Outcome: Serum Bactericidal Assay Using Human Complement Geometric Mean Titers: Groups 1, 2, 3, 4, 6, and 7 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: Groups 1, 3, 4, and 6: at the age of 13 months; Groups 2 and 7: at the age of 16 months
Population: Booster PPP. Here, 'Number analyzed'=participants with available data for specified categories and '0' in number analyzed field signifies none of the participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49 | 27 | 28
titers (1/dilution)
  Serogroup A- at 13 months of age: number analyzed (Participants) | 59 | 0 | 55 | 46 | 25 | 0
  Serogroup A- at 13 months of age | 58.9 [39.9 to 87.2] |  | 98.2 [66.1 to 145.9] | 151.1 [102.2 to 223.4] | 2.7 [2.1 to 3.4] |
  Serogroup A- at 16 months of age: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup A- at 16 months of age |  | 76.1 [50.5 to 114.7] |  |  |  | 2.8 [2.2 to 3.4]
  Serogroup C- at 13 months of age: number analyzed (Participants) | 59 | 0 | 55 | 46 | 26 | 0
  Serogroup C- at 13 months of age | 271.5 [178.5 to 412.9] |  | 179.9 [112.1 to 288.6] | 641.8 [436.4 to 944.1] | 2.8 [2.1 to 3.5] |
  Serogroup C- at 16 months of age: number analyzed (Participants) | 0 | 65 | 0 | 0 | 0 | 26
  Serogroup C- at 16 months of age |  | 272.9 [188.2 to 395.7] |  |  |  | 2.8 [2.2 to 3.5]
  Serogroup Y- at 13 months of age: number analyzed (Participants) | 59 | 0 | 54 | 46 | 26 | 0
  Serogroup Y- at 13 months of age | 253.0 [171.2 to 373.9] |  | 216.7 [156.3 to 300.3] | 396.3 [278.3 to 564.3] | 2.3 [1.9 to 2.7] |
  Serogroup Y- at 16 months of age: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup Y- at 16 months of age |  | 469.5 [351.2 to 627.6] |  |  |  | 2.3 [1.9 to 2.9]
  Serogroup W-135- at 13 months of age: number analyzed (Participants) | 59 | 0 | 54 | 46 | 25 | 0
  Serogroup W-135- at 13 months of age | 355.7 [244.0 to 518.6] |  | 306.4 [210.9 to 445.1] | 384.5 [267.1 to 553.7] | 2.4 [1.8 to 3.2] |
  Serogroup W-135- at 16 months of age: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  Serogroup W-135- at 16 months of age |  | 685.9 [507.1 to 927.7] |  |  |  | 2.2 [1.8 to 2.6]

10. Primary Outcome: Serum Bactericidal Assay Using Human Complement Geometric Mean Titers: Group 5 - Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC.
Time Frame: At the age of 13 months
Population: Analysis was performed on PPP. Here, 'Number analyzed'=participants with available data for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 62
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 59
  Serogroup A | 13.1 [9.5 to 18.1]
  Serogroup C: number analyzed (Participants) | 61
  Serogroup C | 57.8 [39.9 to 83.6]
  Serogroup Y: number analyzed (Participants) | 61
  Serogroup Y | 6.6 [4.8 to 9.0]
  Serogroup W-135: number analyzed (Participants) | 59
  Serogroup W-135 | 6.5 [4.9 to 8.5]

11. Primary Outcome: Percentage of Participants With ≥4-fold Rise in SBA-HC Titer After the Booster Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-HC. Percentage of participants with ≥4-fold rise in each meningococcal serogroups antibody titer (30 days post booster vaccination) were reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: Groups 1, 3, and 4: 30 days post-vaccination at the age of 12 months (i.e. at the age of 13 months), Group 2: 30 days post-vaccination at the age of 15 months (i.e. at the age of 16 months)
Population: Analysis was performed on booster PPP. Here, 'Number analyzed'=participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Groups 5, 6, and 7, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
percentage of participants
  Serogroup A: number analyzed (Participants) | 56 | 62 | 53 | 44
  Serogroup A | 83.9 [71.7 to 92.4] | 85.5 [74.2 to 93.1] | 84.9 [72.4 to 93.3] | 97.7 [88.0 to 99.9]
  Serogroup C: number analyzed (Participants) | 57 | 64 | 53 | 45
  Serogroup C | 93.0 [83.0 to 98.1] | 95.3 [86.9 to 99.0] | 83.0 [70.2 to 91.9] | 97.8 [88.2 to 99.9]
  Serogroup Y: number analyzed (Participants) | 57 | 63 | 52 | 45
  Serogroup Y | 84.2 [72.1 to 92.5] | 92.1 [82.4 to 97.4] | 82.7 [69.7 to 91.8] | 93.3 [81.7 to 98.6]
  Serogroup W-135: number analyzed (Participants) | 57 | 63 | 52 | 45
  Serogroup W-135 | 94.7 [85.4 to 98.9] | 85.7 [74.6 to 93.3] | 90.4 [79.0 to 96.8] | 86.7 [73.2 to 94.9]

12. Primary Outcome: Geometric Mean Fold Rise (GMFR) in SBA-HC Titer After the Booster Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: as for outcome 9
Time Frame: Groups 1, 3 and 4: 30 days post-vaccination at the age of 12 months (i.e. at the age of 13 months), Group 2: 30 days post-vaccination at the age of 15 months (i.e. at the age of 16 months)
Population: Analysis was performed on booster PPP. Here, 'Number analyzed'=participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Groups 5, 6 and 7, as pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
fold rise
  Serogroup A: number analyzed (Participants) | 56 | 62 | 53 | 44
  Serogroup A | 8.3 [5.8 to 11.8] | 12.0 [8.0 to 18.0] | 16.9 [10.9 to 26.0] | 24.5 [17.4 to 34.5]
  Serogroup C: number analyzed (Participants) | 57 | 64 | 53 | 45
  Serogroup C | 19.2 [13.8 to 26.6] | 21.7 [15.6 to 30.1] | 17.1 [11.1 to 26.3] | 25.0 [18.6 to 33.6]
  Serogroup Y: number analyzed (Participants) | 57 | 63 | 52 | 45
  Serogroup Y | 8.7 [6.2 to 12.2] | 14.3 [10.7 to 19.2] | 10.6 [7.5 to 14.8] | 17.3 [11.8 to 25.4]
  Serogroup W-135: number analyzed (Participants) | 57 | 63 | 52 | 45
  Serogroup W-135 | 12.2 [9.1 to 16.4] | 15.1 [10.6 to 21.7] | 13.1 [9.2 to 18.7] | 16.0 [11.2 to 22.9]

13. Primary Outcome: Percentage of Participants With a Serum Bactericidal Assay Using Baby Rabbit Complement (SBA-BR) Titer ≥1:8 and ≥1:128: Groups 1, 2, 3, 4, 6, and 7 - Primary Series Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Primary series PPP was defined as the PPP which was used for reporting data of time points prior to 12 months of age.
Time Frame: Groups 1, 2, 4, 6, and 7: at the age of 7 months; Group 3: at the age of 5 months
Population: Primary series PPP. Here, 'Number analyzed'=participants with available data for specified categories and '0' in number analyzed field signifies none of participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 78 | 81 | 77 | 61 | 45 | 35
percentage of participants
  Serogroup A- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup A- at 5 months of age: ≥1:8 |  |  | 52.6 [40.8 to 64.2] |  |  |
  Serogroup A- at 5 months of age: ≥1:128: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup A- at 5 months of age: ≥1:128 |  |  | 34.2 [23.7 to 46.0] |  |  |
  Serogroup A- at 7 months of age: ≥1:8: number analyzed (Participants) | 70 | 77 | 0 | 55 | 38 | 35
  Serogroup A- at 7 months of age: ≥1:8 | 50.0 [37.8 to 62.2] | 54.5 [42.8 to 65.9] |  | 43.6 [30.3 to 57.7] | 2.6 [0.1 to 13.8] | 2.9 [0.1 to 14.9]
  Serogroup A- at 7 months of age: ≥1:128: number analyzed (Participants) | 70 | 77 | 0 | 55 | 38 | 35
  Serogroup A- at 7 months of age: ≥1:128 | 31.4 [20.9 to 43.6] | 37.7 [26.9 to 49.4] |  | 21.8 [11.8 to 35.0] | 2.6 [0.1 to 13.8] | 2.9 [0.1 to 14.9]
  Serogroup C- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup C- at 5 months of age: ≥1:8 |  |  | 93.4 [85.3 to 97.8] |  |  |
  Serogroup C- at 5 months of age: ≥1:128: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup C- at 5 months of age: ≥1:128 |  |  | 92.1 [83.6 to 97.0] |  |  |
  Serogroup C- at 7 months of age: ≥1:8: number analyzed (Participants) | 70 | 77 | 0 | 57 | 39 | 35
  Serogroup C- at 7 months of age: ≥1:8 | 95.7 [88.0 to 99.1] | 94.8 [87.2 to 98.6] |  | 91.2 [80.7 to 97.1] | 2.6 [0.1 to 13.5] | 8.6 [1.8 to 23.1]
  Serogroup C- at 7 months of age: ≥1:128: number analyzed (Participants) | 70 | 77 | 0 | 57 | 39 | 35
  Serogroup C- at 7 months of age: ≥1:128 | 94.3 [86.0 to 98.4] | 93.5 [85.5 to 97.9] |  | 80.7 [68.1 to 90.0] | 0.0 [0.0 to 9.0] | 5.7 [0.7 to 19.2]
  Serogroup Y- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup Y- at 5 months of age: ≥1:8 |  |  | 98.7 [92.9 to 100.0] |  |  |
  Serogroup Y- at 5 months of age: ≥1:128: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup Y- at 5 months of age: ≥1:128 |  |  | 81.6 [71.0 to 89.5] |  |  |
  Serogroup Y- at 7 months of age: ≥1:8: number analyzed (Participants) | 71 | 77 | 0 | 56 | 39 | 35
  Serogroup Y- at 7 months of age: ≥1:8 | 97.2 [90.2 to 99.7] | 100.0 [95.3 to 100.0] |  | 82.1 [69.6 to 91.1] | 38.5 [23.4 to 55.4] | 37.1 [21.5 to 55.1]
  Serogroup Y- at 7 months of age: ≥1:128: number analyzed (Participants) | 71 | 77 | 0 | 56 | 39 | 35
  Serogroup Y- at 7 months of age: ≥1:128 | 87.3 [77.3 to 94.0] | 92.2 [83.8 to 97.1] |  | 46.4 [33.0 to 60.3] | 15.4 [5.9 to 30.5] | 17.1 [6.6 to 33.6]
  Serogroup W-135- at 5 months of age: ≥1:8: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup W-135- at 5 months of age: ≥1:8 |  |  | 100.0 [95.3 to 100.0] |  |  |
  Serogroup W-135- at 5 months of age: ≥1:128: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup W-135- at 5 months of age: ≥1:128 |  |  | 96.1 [88.9 to 99.2] |  |  |
  Serogroup W-135- at 7 months of age: ≥1:8: number analyzed (Participants) | 70 | 77 | 0 | 56 | 38 | 35
  Serogroup W-135- at 7 months of age: ≥1:8 | 100.0 [94.9 to 100.0] | 98.7 [93.0 to 100.0] |  | 80.4 [67.6 to 89.8] | 13.2 [4.4 to 28.1] | 14.3 [4.8 to 30.3]
  Serogroup W-135- at 7 months of age: ≥1:128: number analyzed (Participants) | 70 | 77 | 0 | 56 | 38 | 35
  Serogroup W-135- at 7 months of age: ≥1:128 | 97.1 [90.1 to 99.7] | 94.8 [87.2 to 98.6] |  | 66.1 [52.2 to 78.2] | 2.6 [0.1 to 13.8] | 5.7 [0.7 to 19.2]

14. Primary Outcome: Percentage of Participants With SBA-BR Titer ≥1:8 and ≥1:128: Groups 1, 2, 3, 4, 6, and 7 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: Groups 1, 3, 4, and 6: at the age of 13 months; Groups 2 and 7: at the age of 16 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49 | 27 | 28
percentage of participants
  Serogroup A- at 13 months of age ≥1:8: number analyzed (Participants) | 56 | 0 | 51 | 42 | 24 | 0
  Serogroup A- at 13 months of age ≥1:8 | 80.4 [67.6 to 89.8] |  | 96.1 [86.5 to 99.5] | 95.2 [83.8 to 99.4] | 8.3 [1.0 to 27.0] |
  Serogroup A- at 13 months of age ≥1:128: number analyzed (Participants) | 56 | 0 | 51 | 42 | 24 | 0
  Serogroup A- at 13 months of age ≥1:128 | 69.6 [55.9 to 81.2] |  | 88.2 [76.1 to 95.6] | 90.5 [77.4 to 97.3] | 4.2 [0.1 to 21.1] |
  Serogroup A- at 16 months of age ≥1:8: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup A- at 16 months of age ≥1:8 |  | 81.4 [69.1 to 90.3] |  |  |  | 0.0 [0.0 to 14.8]
  Serogroup A- at 16 months of age ≥1:128: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup A- at 16 months of age ≥1:128 |  | 74.6 [61.6 to 85.0] |  |  |  | 0.0 [0.0 to 14.8]
  Serogroup C- at 13 months of age ≥1:8: number analyzed (Participants) | 57 | 0 | 53 | 43 | 24 | 0
  Serogroup C- at 13 months of age ≥1:8 | 93.0 [83.0 to 98.1] |  | 88.7 [77.0 to 95.7] | 100.0 [91.8 to 100.0] | 16.7 [4.7 to 37.4] |
  Serogroup C- at 13 months of age ≥1:128: number analyzed (Participants) | 57 | 0 | 53 | 43 | 24 | 0
  Serogroup C- at 13 months of age ≥1:128 | 93.0 [83.0 to 98.1] |  | 86.8 [74.7 to 94.5] | 97.7 [87.7 to 99.9] | 16.7 [4.7 to 37.4] |
  Serogroup C- at 16 months of age ≥1:8: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 24
  Serogroup C- at 16 months of age ≥1:8 |  | 98.3 [90.9 to 100.0] |  |  |  | 8.3 [1.0 to 27.0]
  Serogroup C- at 16 months of age ≥1:128: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 24
  Serogroup C- at 16 months of age ≥1:128 |  | 96.6 [88.3 to 96.6] |  |  |  | 0.0 [0.0 to 14.2]
  Serogroup Y- at 13 months of age ≥1:8: number analyzed (Participants) | 56 | 0 | 52 | 42 | 24 | 0
  Serogroup Y- at 13 months of age ≥1:8 | 100.0 [93.6 to 100.0] |  | 100.0 [93.2 to 100.0] | 100.0 [91.6 to 100.0] | 66.7 [44.7 to 84.4] |
  Serogroup Y- at 13 months of age ≥1:128: number analyzed (Participants) | 56 | 0 | 52 | 42 | 24 | 0
  Serogroup Y- at 13 months of age ≥1:128 | 94.6 [85.1 to 98.9] |  | 94.2 [84.1 to 98.8] | 100.0 [91.6 to 100.0] | 37.5 [18.8 to 59.4] |
  Serogroup Y- at 16 months of age ≥1:8: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup Y- at 16 months of age ≥1:8 |  | 100.0 [93.9 to 100.0] |  |  |  | 73.9 [51.6 to 89.8]
  Serogroup Y- at 16 months of age ≥1:128: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup Y- at 16 months of age ≥1:128 |  | 96.6 [88.3 to 99.6] |  |  |  | 30.4 [13.2 to 52.9]
  Serogroup W-135- at 13 months of age ≥1:8: number analyzed (Participants) | 55 | 0 | 51 | 42 | 24 | 0
  Serogroup W-135- at 13 months of age ≥1:8 | 100.0 [93.5 to 100.0] |  | 98.0 [89.6 to 100.0] | 97.6 [87.4 to 99.9] | 16.7 [4.7 to 37.4] |
  Serogroup W-135- at 13 months of age ≥1:128: number analyzed (Participants) | 55 | 0 | 51 | 42 | 24 | 0
  Serogroup W-135- at 13 months of age ≥1:128 | 98.2 [90.3 to 100.0] |  | 94.1 [83.8 to 98.8] | 95.2 [83.8 to 99.4] | 0.0 [0.0 to 14.2] |
  Serogroup W-135- at 16 months of age ≥1:8: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup W-135- at 16 months of age ≥1:8 |  | 100.0 [93.9 to 100.0] |  |  |  | 17.4 [5.0 to 38.8]
  Serogroup W-135- at 16 months of age ≥1:128: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup W-135- at 16 months of age ≥1:128 |  | 98.3 [90.9 to 100.0] |  |  |  | 4.3 [0.1 to 21.9]

15. Primary Outcome: Percentage of Participants With SBA-BR Titer ≥1:8 and ≥1:128: Group 5 - Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR.
Time Frame: At the age of 13 months
Population: Analysis was performed on PPP. Here, 'Overall number of participant analyzed'=participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 58
percentage of participants
  Serogroup A: ≥1:8 | 62.1 [48.4 to 74.5]
  Serogroup A: ≥1:128 | 46.6 [33.3 to 60.1]
  Serogroup C: ≥1:8 | 91.4 [81.0 to 97.1]
  Serogroup C: ≥1:128 | 82.8 [70.6 to 91.4]
  Serogroup Y: ≥1:8 | 94.8 [85.6 to 98.9]
  Serogroup Y: ≥1:128 | 70.7 [57.3 to 81.9]
  Serogroup W-135: ≥1:8 | 100.0 [93.8 to 100.0]
  Serogroup W-135: ≥1:128 | 86.2 [74.6 to 93.9]

16. Primary Outcome: Percentage of Participants With SBA-BR Pre-Booster Titer ≥1:8 Who Then Achieved ≥4-Fold Rise in SBA-BR Titer After Booster Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Pre-booster titer was defined as titer value reported before the age of 12 months. Percentage of participants whose pre-booster titer was ≥1:8 and achieved ≥4-fold rise in each meningococcal serogroups antibody titer (30 days post booster vaccination) were reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
percentage of participants
  Serogroup A: number analyzed (Participants) | 3 | 5 | 6 | 6
  Serogroup A | 100.0 [29.2 to 100.0] | 100.0 [47.8 to 100.0] | 33.3 [4.3 to 77.7] | 66.7 [22.3 to 95.7]
  Serogroup C: number analyzed (Participants) | 29 | 22 | 22 | 28
  Serogroup C | 86.2 [68.3 to 96.1] | 86.4 [65.1 to 97.1] | 77.3 [54.6 to 92.2] | 96.4 [81.7 to 99.9]
  Serogroup Y: number analyzed (Participants) | 50 | 47 | 48 | 36
  Serogroup Y | 70.0 [55.4 to 82.1] | 83.0 [69.2 to 92.4] | 81.3 [67.4 to 91.1] | 77.8 [60.8 to 89.9]
  Serogroup W-135: number analyzed (Participants) | 47 | 47 | 35 | 31
  Serogroup W-135 | 85.1 [71.7 to 93.8] | 87.2 [74.3 to 95.2] | 82.9 [66.4 to 93.4] | 80.6 [62.5 to 92.5]

17. Primary Outcome: Percentage of Participants With SBA-BR Pre-Vaccination Titer ≥1:8 Who Then Achieved ≥4-Fold Rise in SBA-BR Titer After Vaccination: Group 5 - Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Percentage of participants whose pre-vaccination titer was ≥1:8 and achieved ≥4-fold rise in each meningococcal serogroups antibody titer at the age of Month 13 (i.e. 30-days post vaccination at Month 12) were reported.
Time Frame: 30 days post-vaccination at the age of 12 months (i.e. at the age of 13 months)
Population: Analysis was performed on PPP. Here, 'Overall number of participants analyzed= participants evaluable for this outcome measure' and 'Number analyzed'=participants with available data for specified category. In addition, '0' in number analyzed field signifies none of the participants had titer ≥1:8.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 30
percentage of participants
  Serogroup A: number analyzed (Participants) | 0
  Serogroup C: number analyzed (Participants) | 3
  Serogroup C | 66.7 [9.4 to 99.2]
  Serogroup Y | 53.3 [34.3 to 71.7]
  Serogroup W-135: number analyzed (Participants) | 15
  Serogroup W-135 | 93.3 [68.1 to 99.8]

18. Primary Outcome: Percentage of Participants With SBA-BR Pre-Booster Titer <1:8 Who Then Achieved ≥4-Fold Rise in SBA-BR Titers After Booster Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Pre-booster titer was defined as titer value reported before the age of 12 months. Percentage of participants whose pre-booster titer was <1:8 and achieved ≥4-fold rise in each meningococcal serogroups antibody titer (30-days post booster vaccination) were reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
percentage of participants
  Serogroup A: number analyzed (Participants) | 50 | 48 | 44 | 32
  Serogroup A | 78.0 [64.0 to 88.5] | 79.2 [65.0 to 89.5] | 95.5 [84.5 to 99.4] | 93.8 [79.2 to 99.2]
  Serogroup C: number analyzed (Participants) | 25 | 31 | 30 | 12
  Serogroup C | 88.0 [68.8 to 97.5] | 96.8 [83.3 to 99.9] | 83.3 [65.3 to 94.4] | 100.0 [73.5 to 100.0]
  Serogroup Y: number analyzed (Participants) | 3 | 6 | 3 | 2
  Serogroup Y | 100.0 [29.2 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [15.8 to 100.0]
  Serogroup W-135: number analyzed (Participants) | 5 | 6 | 15 | 7
  Serogroup W-135 | 100.0 [47.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [78.2 to 100.0] | 85.7 [42.1 to 99.6]

19. Primary Outcome: Percentage of Participants With SBA-BR Pre-Vaccination Titer <1:8 Who Then Achieved ≥4-Fold Rise in SBA-BR Titer After Vaccination: Group 5 - Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Pre-vaccination titer was defined as titer value reported before the age of 12 months. Percentage of participants with pre-vaccination titer <1:8 and who achieved ≥4-fold rise in each meningococcal serogroups antibody titer (30 days post-vaccination) were reported.
Time Frame: 30 days post-vaccination at the age of 12 months (i.e. at the age of 13 months)
Population: Analysis was performed on PPP. Here, 'Number analyzed'=participants with available data for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 62
percentage of participants
  Serogroup A: number analyzed (Participants) | 55
  Serogroup A | 61.8 [47.7 to 74.6]
  Serogroup C: number analyzed (Participants) | 54
  Serogroup C | 90.7 [79.7 to 96.9]
  Serogroup Y: number analyzed (Participants) | 27
  Serogroup Y | 74.1 [53.7 to 88.9]
  Serogroup W-135: number analyzed (Participants) | 42
  Serogroup W-135 | 97.6 [87.4 to 99.9]

20. Primary Outcome: Percentage of Participants With ≥4-fold Rise in SBA-BR Titer After the Booster Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Percentage of participants with ≥4-fold rise in each meningococcal serogroups antibody titer (30-days post booster vaccination) were reported. Booster PPP was defined as the PPP which was used for reporting data of time points at and after the age of 12 months.
Time Frame: Groups 1, 3, and 4: 30 days post booster vaccination (i.e., at the age of 13 months); Group 2: 30 days post booster vaccination (i.e., at the age of 16 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
percentage of participants
  Serogroup A: number analyzed (Participants) | 53 | 53 | 50 | 38
  Serogroup A | 79.2 [65.9 to 89.2] | 81.1 [68.0 to 90.6] | 88.0 [75.7 to 95.5] | 89.5 [75.2 to 97.1]
  Serogroup C: number analyzed (Participants) | 54 | 53 | 52 | 40
  Serogroup C | 87.0 [75.1 to 94.6] | 92.5 [81.8 to 97.9] | 80.8 [67.5 to 90.4] | 97.5 [86.8 to 99.9]
  Serogroup Y: number analyzed (Participants) | 53 | 53 | 51 | 38
  Serogroup Y | 71.7 [57.7 to 83.2] | 84.9 [72.4 to 93.3] | 82.4 [69.1 to 91.6] | 78.9 [62.7 to 90.4]
  Serogroup W-135: number analyzed (Participants) | 52 | 53 | 50 | 38
  Serogroup W-135 | 86.5 [74.2 to 94.4] | 88.7 [77.0 to 95.7] | 88.0 [75.7 to 95.5] | 81.6 [65.7 to 92.3]

21. Primary Outcome: Serum Bactericidal Assay Using Baby Rabbit Complement Geometric Mean Titers: Groups 1, 2, 3, 4, 6, and 7 - Primary Series Per-Protocol Population
Description: as for outcome 13
Time Frame: Groups 1, 2, 4, 6, and 7: at the age of 7 months; Group 3: at the age of 5 months
Population: Primary series PPP. 'Number analyzed'=participants with available data for specified categories and '0' in number analyzed field signifies none of the participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 78 | 81 | 77 | 61 | 45 | 35
titers (1/dilution)
  Serogroup A- at 5 months of age: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup A- at 5 months of age |  |  | 26.2 [16.6 to 41.4] |  |  |
  Serogroup A- at 7 months of age: number analyzed (Participants) | 70 | 77 | 0 | 55 | 38 | 35
  Serogroup A- at 7 months of age | 24.0 [15.0 to 38.5] | 27.5 [17.8 to 42.3] |  | 17.7 [10.9 to 28.6] | 4.4 [3.6 to 5.3] | 4.6 [3.5 to 6.1]
  Serogroup C- at 5 months of age: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup C- at 5 months of age |  |  | 807.8 [550.2 to 1186.1] |  |  |
  Serogroup C- at 7 months of age: number analyzed (Participants) | 70 | 77 | 0 | 57 | 39 | 35
  Serogroup C- at 7 months of age | 696.0 [489.4 to 989.8] | 689.1 [478.4 to 992.6] |  | 377.8 [231.1 to 617.6] | 4.3 [3.7 to 5.0] | 5.4 [3.8 to 7.7]
  Serogroup Y- at 5 months of age: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup Y- at 5 months of age |  |  | 265.5 [198.2 to 355.7] |  |  |
  Serogroup Y- at 7 months of age: number analyzed (Participants) | 71 | 77 | 0 | 56 | 39 | 35
  Serogroup Y- at 7 months of age | 333.2 [239.6 to 463.4] | 530.8 [420.7 to 669.6] |  | 53.2 [34.5 to 81.8] | 12.3 [7.4 to 20.2] | 13.1 [7.1 to 24.2]
  Serogroup W-135- at 5 months of age: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  Serogroup W-135- at 5 months of age |  |  | 526.2 [417.3 to 663.6] |  |  |
  Serogroup W-135- at 7 months of age: number analyzed (Participants) | 70 | 77 | 0 | 56 | 38 | 35
  Serogroup W-135- at 7 months of age | 655.8 [511.5 to 840.9] | 781.7 [595.1 to 1026.7] |  | 120.3 [68.8 to 210.4] | 5.9 [4.0 to 8.7] | 5.9 [4.1 to 8.5]

22. Primary Outcome: Serum Bactericidal Assay Using Baby Rabbit Complement Geometric Mean Titers: Groups 1, 2, 3, 4, 6, and 7 - Booster Per-Protocol Population
Description: as for outcome 14
Time Frame: Groups 1, 3, 4, and 6: at the age of 13 months; Group 2 and 7: at the age of 16 months
Population: Booster PPP. Here, 'Number analyzed'=participants with available data for specified categories and '0' in number analyzed field signifies none of participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in timeframe and pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49 | 27 | 28
titers (1/dilution)
  Serogroup A- at 13 months of age: number analyzed (Participants) | 56 | 0 | 51 | 42 | 24 | 0
  Serogroup A- at 13 months of age | 137.9 [79.8 to 238.2] |  | 256.0 [183.5 to 357.2] | 406.4 [256.1 to 644.8] | 5.3 [3.5 to 8.1] |
  Serogroup A- at 16 months of age: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup A- at 16 months of age |  | 169.7 [100.8 to 285.7] |  |  |  | 4.0 [NA to NA] — Here, 'NA' signifies that 95% confidence interval was not computable as the standard deviation of the sample was 0, since all subjects had the same value.
  Serogroup C- at 13 months of age: number analyzed (Participants) | 57 | 0 | 53 | 43 | 24 | 0
  Serogroup C- at 13 months of age | 975.4 [606.5 to 1568.6] |  | 691.7 [387.3 to 1235.2] | 3164.8 [2149.8 to 4659.2] | 7.3 [4.1 to 13.2] |
  Serogroup C- at 16 months of age: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 24
  Serogroup C- at 16 months of age |  | 1086.0 [766.0 to 1539.6] |  |  |  | 4.8 [3.7 to 6.1]
  Serogroup Y- at 13 months of age: number analyzed (Participants) | 56 | 0 | 52 | 42 | 24 | 0
  Serogroup Y- at 13 months of age | 579.5 [444.5 to 755.4] |  | 642.2 [471.1 to 875.4] | 942.9 [707.6 to 1256.4] | 32.9 [15.8 to 68.7] |
  Serogroup Y- at 16 months of age: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 23
  Serogroup Y- at 16 months of age |  | 1024.0 [778.1 to 1347.5] |  |  |  | 43.3 [21.1 to 88.5]
  Serogroup W-135- at 13 months of age: number analyzed (Participants) | 55 | 0 | 51 | 42 | 24 | 0
  Serogroup W-135- at 13 months of age | 1011.2 [763.9 to 1338.6] |  | 769.7 [532.6 to 1112.4] | 826.3 [570.1 to 1197.5] | 5.8 [4.0 to 8.5] |
  Serogroup W-135- at 16 months of age: number analyzed (Participants) | 0 | 59 | 0 | 0 | 0 | 28
  Serogroup W-135- at 16 months of age |  | 1389.8 [1027.1 to 1880.5] |  |  |  | 6.3 [3.9 to 10.1]

23. Primary Outcome: Serum Bactericidal Assay Using Baby Rabbit Complement Geometric Mean Titers in Group 5: Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR.
Time Frame: At the age of 13 months
Population: Analysis was performed on PPP. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 58
titers (1/dilution)
  Serogroup A | 42.6 [25.2 to 72.1]
  Serogroup C | 403.1 [247.7 to 656.1]
  Serogroup Y | 166.5 [109.5 to 253.2]
  Serogroup W-135 | 403.1 [288.3 to 563.8]

24. Primary Outcome: Geometric Mean Fold Rise in Serum Bactericidal Assay Using Baby Rabbit Complement Titer After the Booster Vaccination: Groups 1, 2, 3, and 4 - Booster Per-Protocol Population
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR. Percentage of participants with GMFR in each meningococcal serogroups antibody titer (30-days post booster vaccination) were reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: Groups 1, 3, and 4: 30 days post booster vaccination at the age of 12 months (i.e., at the age of 13 months); Group 2: 30 days post booster vaccination at the age of 15 months (i.e. at the age of 16 months)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months
Number analyzed (Participants) | 65 | 68 | 57 | 49
fold rise
  Serogroup A: number analyzed (Participants) | 53 | 53 | 50 | 38
  Serogroup A | 15.8 [9.6 to 26.0] | 21.1 [13.0 to 34.1] | 22.3 [15.0 to 33.3] | 32.6 [19.8 to 53.6]
  Serogroup C: number analyzed (Participants) | 54 | 53 | 52 | 40
  Serogroup C | 26.7 [16.3 to 43.8] | 37.9 [24.2 to 59.5] | 27.3 [15.3 to 48.7] | 32.0 [18.8 to 54.6]
  Serogroup Y: number analyzed (Participants) | 53 | 53 | 51 | 38
  Serogroup Y | 6.1 [4.2 to 8.7] | 10.0 [6.5 to 15.3] | 7.1 [4.8 to 10.4] | 8.6 [5.5 to 13.4]
  Serogroup W-135: number analyzed (Participants) | 52 | 53 | 50 | 38
  Serogroup W-135 | 10.2 [7.2 to 14.3] | 12.8 [9.1 to 18.1] | 19.7 [12.1 to 32.0] | 11.1 [7.2 to 17.1]

25. Primary Outcome: Antibody Titer/Concentration to All the Antigens Contained in Pentacel Vaccines: Groups 1, 2, 4, 6, and 7 - Primary Series Per-Protocol Population
Description: Pentacel vaccine is Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined). Antibody titer to all antigens contained in pentacel vaccines (i.e., Anti-PRP, Anti-Diptheria, Anti-pertussis [pertussis toxoid [PT], pertactin [PRN], filamentous hemagglutinin [FHA], and fimbriae [FIM]], Anti-poliovirus [anti-poliovirus Type 1, Type 2 and Type 3] and anti-tetanus) were reported. Primary series PPP was defined as the PPP which was used for reporting data of time points prior to 12 months of age.
Time Frame: At the age of 7 months
Population: Analysis was performed on primary series PPP. Here, 'Number analyzed'=participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 5, as pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 78 | 81 | 61 | 45 | 35
titers (1/dilution)
  Anti-PRP: number analyzed (Participants) | 38 | 47 | 32 | 26 | 21
  Anti-PRP | 4.1 [2.3 to 7.1] | 3.8 [2.1 to 6.6] | 3.2 [2.0 to 5.3] | 5.4 [3.1 to 9.2] | 3.8 [1.5 to 9.4]
  Anti-Diphtheria: number analyzed (Participants) | 37 | 44 | 32 | 24 | 21
  Anti-Diphtheria | 0.3 [0.3 to 0.5] | 0.6 [0.4 to 0.8] | 0.6 [0.4 to 0.9] | 0.6 [0.4 to 0.8] | 0.6 [0.4 to 1.0]
  PT: number analyzed (Participants) | 37 | 46 | 32 | 24 | 21
  PT | 65.0 [51.7 to 81.6] | 66.8 [53.2 to 83.7] | 60.5 [49.7 to 73.7] | 61.4 [45.8 to 82.5] | 79.2 [61.9 to 101.3]
  FHA: number analyzed (Participants) | 37 | 46 | 32 | 24 | 21
  FHA | 67.2 [54.4 to 83.0] | 81.6 [67.2 to 98.9] | 69.6 [52.8 to 91.9] | 60.9 [47.2 to 78.7] | 93.2 [70.5 to 123.0]
  PRN: number analyzed (Participants) | 37 | 46 | 32 | 24 | 21
  PRN | 31.9 [21.3 to 47.7] | 33.7 [24.0 to 47.2] | 36.7 [25.0 to 53.9] | 34.5 [21.6 to 55.1] | 52.0 [29.6 to 91.4]
  FIM: number analyzed (Participants) | 37 | 45 | 32 | 24 | 21
  FIM | 154.8 [110.7 to 216.5] | 177.5 [122.3 to 257.6] | 186.8 [117.4 to 297.3] | 194.0 [137.0 to 274.8] | 194.4 [111.8 to 338.3]
  Anti-Poliovirus Type 1: number analyzed (Participants) | 36 | 44 | 32 | 23 | 21
  Anti-Poliovirus Type 1 | 273.9 [157.6 to 476.0] | 696.1 [464.1 to 1044.1] | 716.2 [381.0 to 1346.5] | 543.9 [303.5 to 974.5] | 327.9 [165.4 to 650.0]
  Anti-Poliovirus Type 2: number analyzed (Participants) | 36 | 44 | 32 | 24 | 21
  Anti-Poliovirus Type 2 | 886.3 [604.5 to 1299.5] | 1494.5 [1041.3 to 2145.0] | 1401.8 [896.5 to 2192.0] | 1054.0 [639.7 to 1736.7] | 1075.9 [550.6 to 2102.4]
  Anti-Poliovirus Type 3: number analyzed (Participants) | 37 | 44 | 31 | 24 | 21
  Anti-Poliovirus Type 3 | 968.0 [606.6 to 1544.8] | 1381.4 [845.1 to 2257.9] | 1674.7 [962.4 to 2914.0] | 1069.3 [689.6 to 1658.1] | 927.5 [469.7 to 1831.9]
  Anti-tetanus: number analyzed (Participants) | 73 | 81 | 59 | 44 | 35
  Anti-tetanus | 1.7 [1.4 to 2.0] | 1.9 [1.6 to 2.2] | 1.6 [1.3 to 2.0] | 1.3 [1.1 to 1.7] | 1.5 [1.1 to 1.9]

26. Primary Outcome: Antibody Titer/Concentration to All Antigens Contained in Pentacel Vaccines: Groups 2 and 7 - Booster Per-Protocol Population
Description: Pentacel vaccine is Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate) Vaccine Combined (DTaP-IPV/Hib combined). Antibody titer to all antigens contained in pentacel vaccines (i.e., Anti-PRP, Anti-Diptheria, Anti-pertussis [PT, PRN, FHA, and FIM], Anti-poliovirus [anti-poliovirus Type 1, Type 2, and Type 3], and Anti-tetanus) were reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: At the age of 16 months
Population: Booster PPP. Here, 'Number analyzed'=participants with available data for specified categories. Data for this outcome measure was not planned to be collected and analyzed for Groups 1, 3, 4, 5, and 6, as pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 68 | 28
titers (1/dilution)
  Anti-PRP: number analyzed (Participants) | 60 | 25
  Anti-PRP | 17.2 [12.7 to 23.4] | 18.0 [8.4 to 38.7]
  Anti-Diphtheria: number analyzed (Participants) | 61 | 25
  Anti-Diphtheria | 5.3 [4.3 to 6.5] | 5.6 [4.2 to 7.3]
  PT: number analyzed (Participants) | 63 | 26
  PT | 108.6 [89.5 to 131.7] | 102.6 [80.5 to 130.7]
  FHA: number analyzed (Participants) | 63 | 26
  FHA | 134.0 [108.3 to 165.9] | 122.5 [91.8 to 163.3]
  PRN: number analyzed (Participants) | 63 | 26
  PRN | 155.4 [112.8 to 214.2] | 122.0 [75.9 to 196.0]
  FIM: number analyzed (Participants) | 61 | 25
  FIM | 484.7 [376.1 to 624.6] | 619.3 [404.0 to 949.3]
  Anti-Poliovirus Type 1: number analyzed (Participants) | 61 | 24
  Anti-Poliovirus Type 1 | 2498.6 [1900.1 to 3285.5] | 1625.6 [853.8 to 3094.9]
  Anti-Poliovirus Type 2: number analyzed (Participants) | 61 | 24
  Anti-Poliovirus Type 2 | 3718.9 [2922.5 to 4732.3] | 3756.1 [2344.6 to 6017.2]
  Anti-Poliovirus Type 3: number analyzed (Participants) | 61 | 24
  Anti-Poliovirus Type 3 | 3473.8 [2546.0 to 4739.6] | 2733.8 [1638.6 to 4560.8]
  Anti-tetanus: number analyzed (Participants) | 64 | 26
  Anti-tetanus | 5.1 [4.1 to 6.3] | 2.7 [2.0 to 3.6]

27. Primary Outcome: Percentage of Participants With Antibody Concentration ≥0.35 μg/mL for Serotypes in Prevnar 7 or 13 Vaccine: Groups 1, 2, 4, 6, and 7 - Primary Series Per-Protocol Population
Description: Percentage of participants with anti-pneumococcal antibody concentrations ≥0.35 μg/mL for serotypes in Prevnar 7 or 13 vaccine i.e. 4, 6B, 9V, 14, 18C, 19F, and 23F is reported. Primary series PPP was defined as the PPP which was used for reporting data of time points prior to 12 months of age.
Time Frame: At the age of 7 months
Population: Analysis was performed on primary series PPP. Here, 'Number analyzed'=participants with available data for specified categories. Data for this outcome measure was not planned to be collected and analyzed for Group 3, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 78 | 81 | 61 | 45 | 35
percentage of participants
  Serotype 4: ≥0.35 μg/mL: number analyzed (Participants) | 36 | 34 | 23 | 18 | 14
  Serotype 4: ≥0.35 μg/mL | 100.0 [90.3 to 100.0] | 100.0 [89.7 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [81.5 to 100.0] | 92.9 [66.1 to 99.8]
  Serotype 6B: ≥0.35 μg/mL: number analyzed (Participants) | 35 | 34 | 23 | 18 | 14
  Serotype 6B: ≥0.35 μg/mL | 94.3 [80.8 to 99.3] | 91.2 [76.3 to 98.1] | 82.6 [61.2 to 95.0] | 77.8 [52.4 to 93.6] | 92.9 [66.1 to 99.8]
  Serotype 9V: ≥0.35 μg/mL: number analyzed (Participants) | 36 | 34 | 23 | 18 | 14
  Serotype 9V: ≥0.35 μg/mL | 97.2 [85.5 to 99.9] | 100.0 [89.7 to 100.0] | 95.7 [78.1 to 99.9] | 94.4 [72.7 to 99.9] | 85.7 [57.2 to 98.2]
  Serotype 14: ≥0.35 μg/mL: number analyzed (Participants) | 36 | 34 | 23 | 18 | 14
  Serotype 14: ≥0.35 μg/mL | 100.0 [90.3 to 100.0] | 100.0 [89.7 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [81.5 to 100.0] | 100.0 [76.8 to 100.0]
  Serotype 18C: ≥0.35 μg/mL: number analyzed (Participants) | 35 | 34 | 23 | 18 | 14
  Serotype 18C: ≥0.35 μg/mL | 97.1 [85.1 to 99.9] | 100.0 [89.7 to 100.0] | 95.7 [78.1 to 99.9] | 100.0 [81.5 to 100.0] | 100.0 [76.8 to 100.0]
  Serotype 19F: ≥0.35 μg/mL: number analyzed (Participants) | 36 | 34 | 23 | 18 | 14
  Serotype 19F: ≥0.35 μg/mL | 97.2 [85.5 to 99.9] | 100.0 [89.7 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [81.5 to 100.0] | 100.0 [76.8 to 100.0]
  Serotype 23F: ≥0.35 μg/mL: number analyzed (Participants) | 36 | 34 | 23 | 18 | 14
  Serotype 23F: ≥0.35 μg/mL | 94.4 [81.3 to 99.3] | 97.1 [84.7 to 99.9] | 91.3 [72.0 to 98.9] | 83.3 [58.6 to 96.4] | 92.9 [66.1 to 99.8]

28. Primary Outcome: Percentage of Participants With Antibody Concentration ≥0.35 μg/mL and ≥1.0 μg/mL for Serotypes in Prevnar 7 or 13 Vaccine: Groups 1, 3, 4, and 6 - Booster Series Per-Protocol Population
Description: Percentage of participants with anti-pneumococcal antibody concentrations ≥0.35 μg/mL and ≥1.0 μg/mL for serotypes in Prevnar 7 or 13 vaccine i.e. 4, 6B, 9V, 14, 18C, 19F and 23F is reported. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: At the age of 13 months
Population: Analysis was performed on booster PPP. Here, 'Number analyzed'=participants with available data for specified categories. Data for this outcome measure was not planned to be collected and analyzed for Groups 2 and 7.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months
Number analyzed (Participants) | 65 | 57 | 49 | 27
percentage of participants
  Serotype 4: ≥0.35 μg/mL: number analyzed (Participants) | 25 | 21 | 2 | 10
  Serotype 4: ≥0.35 μg/mL | 96.0 [79.6 to 99.9] | 100.0 [83.9 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [69.2 to 100.0]
  Serotype 6B: ≥0.35 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 6B: ≥0.35 μg/mL | 100.0 [86.3 to 100.0] | 100.0 [83.9 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [69.2 to 100.0]
  Serotype 9V: ≥0.35 μg/mL: number analyzed (Participants) | 25 | 21 | 18 | 10
  Serotype 9V: ≥0.35 μg/mL | 96.0 [79.6 to 99.9] | 100.0 [83.9 to 100.0] | 100.0 [81.5 to 100.0] | 100.0 [69.2 to 100.0]
  Serotype 14: ≥0.35 μg/mL: number analyzed (Participants) | 25 | 20 | 19 | 10
  Serotype 14: ≥0.35 μg/mL | 100.0 [86.3 to 100.0] | 100.0 [83.2 to 100.0] | 100.0 [82.4 to 100.0] | 90.0 [55.5 to 99.7]
  Serotype 18C: ≥0.35 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 18C: ≥0.35 μg/mL | 100.0 [86.3 to 100.0] | 100.0 [83.9 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [69.2 to 100.0]
  Serotype 19F: ≥0.35 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 19F: ≥0.35 μg/mL | 100.0 [86.3 to 100.0] | 100.0 [83.9 to 100.0] | 94.7 [74.0 to 99.9] | 100.0 [69.2 to 100.0]
  Serotype 23F: ≥0.35 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 23F: ≥0.35 μg/mL | 100.0 [86.3 to 100.0] | 100.0 [83.9 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [69.2 to 100.0]
  Serotype 4: ≥1.0 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 4: ≥1.0 μg/mL | 80.0 [59.3 to 93.2] | 66.7 [43.0 to 85.4] | 84.2 [60.4 to 96.6] | 60.0 [26.2 to 87.8]
  Serotype 6B: ≥1.0 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 6B: ≥1.0 μg/mL | 96.0 [79.6 to 99.9] | 100.0 [83.9 to 100.0] | 100.0 [82.4 to 100.0] | 90.0 [55.5 to 99.7]
  Serotype 9V: ≥1.0 μg/mL: number analyzed (Participants) | 25 | 21 | 18 | 10
  Serotype 9V: ≥1.0 μg/mL | 84.0 [63.9 to 95.5] | 76.2 [52.8 to 91.8] | 77.8 [52.4 to 93.6] | 60.0 [26.2 to 87.8]
  Serotype 14: ≥1.0 μg/mL: number analyzed (Participants) | 25 | 20 | 19 | 10
  Serotype 14: ≥1.0 μg/mL | 100.0 [86.3 to 100.0] | 100.0 [83.2 to 100.0] | 100.0 [82.4 to 100.0] | 90.0 [55.5 to 99.7]
  Serotype 18C: ≥1.0 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 18C: ≥1.0 μg/mL | 88.0 [68.8 to 97.5] | 85.7 [63.7 to 97.0] | 89.5 [66.9 to 98.7] | 70.0 [34.8 to 93.3]
  Serotype 19F: ≥1.0 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 19F: ≥1.0 μg/mL | 96.0 [79.6 to 99.9] | 95.2 [76.2 to 99.9] | 94.7 [74.0 to 99.9] | 100.0 [69.2 to 100.0]
  Serotype 23F: ≥1.0 μg/mL: number analyzed (Participants) | 25 | 21 | 19 | 10
  Serotype 23F: ≥1.0 μg/mL | 100.0 [86.3 to 100.0] | 90.5 [69.6 to 98.8] | 89.5 [66.9 to 98.7] | 90.0 [55.5 to 99.7]

29. Primary Outcome: Percentage of Participants With Antibody Concentration ≥0.35 μg/mL and ≥1.0 μg/mL for Serotypes in Prevnar 7 or 13 Vaccine: Group 5- Per-Protocol Population
Description: Percentage of participants with anti-pneumococcal antibody concentrations ≥0.35 μg/mL and ≥1.0 μg/mL for serotypes in Prevnar 7 or 13 vaccine i.e. 4, 6B, 9V, 14, 18C, 19F and 23F is reported.
Time Frame: At the age of 13 months
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 12
percentage of participants
  Serotype 4: ≥0.35 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 6B: ≥0.35 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 9V: ≥0.35 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 14: ≥0.35 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 18C: ≥0.35 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 19F: ≥0.35 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 23F: ≥0.35 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 4: ≥1.0 μg/mL | 66.7 [34.9 to 90.1]
  Serotype 6B: ≥1.0 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 9V: ≥1.0 μg/mL | 91.7 [61.5 to 99.8]
  Serotype 14: ≥1.0 μg/mL | 100.0 [73.5 to 100.0]
  Serotype 18C: ≥1.0 μg/mL | 75.0 [42.8 to 94.5]
  Serotype 19F: ≥1.0 μg/mL | 83.3 [51.6 to 97.9]
  Serotype 23F: ≥1.0 μg/mL | 91.7 [61.5 to 99.8]

30. Primary Outcome: Percentage of Participants With Antibodies to All Antigens Contained in M-M-RII and VARIVAX Vaccines: Groups 1 and 6 - Booster Per-Protocol Population
Description: Antibodies responses were measured by ELISA. Antigens contained in M-M-RII: Measles, Mumps, and Rubella and in Varivax®: Varicella. Percentage of participants with anti-measles, anti-mumps, anti-rubella, and anti-varicella antibody concentration that met the respective mentioned criterion were reported: Measles: ≥255 milli-International Units per milliliter (mIU/mL); Mumps: ≥10 Antibody units per milliliter (AbU/mL); Rubella: ≥10 International Units per milliliter (IU/mL); Varicella: ≥5 glycoprotein based enzyme-linked immunosorbent assay (gpELISA) unit/mL. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months.
Time Frame: At the age of 13 months
Population: Analysis was performed on booster PPP. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Groups 2, 3, 4, 5, and 7, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months
Number analyzed (Participants) | 31 | 14
percentage of participants
  Measles: ≥255 mIU/mL | 100.0 [88.8 to 100.0] | 100.0 [76.8 to 100.0]
  Mumps: ≥10 AbU/mL | 100.0 [88.8 to 100.0] | 100.0 [76.8 to 100.0]
  Rubella: ≥10 IU/mL | 100.0 [88.8 to 100.0] | 100.0 [76.8 to 100.0]
  Varicella: ≥5 gpELISA unit/mL | 100.0 [88.8 to 100.0] | 100.0 [76.8 to 100.0]

31. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibody Titers to Tetanus Toxoid: Groups 1, 2, 3, 4, 6, and 7 - Primary Series Per-Protocol Population
Description: Antibody concentrations against tetanus toxoid were measured by ELISA and expressed as GMC. Primary series PPP was defined as the PPP which was used for reporting data of time points prior to 12 months of age. Here, '0' in number analyzed field signifies none of the participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Time Frame: Groups 1, 2, 4, 6, and 7: at the age of 7 months; Group 3: at the age of 5 months
Population: Analysis was performed on Primary series PPP. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure and 'Number analyzed'=participants with available data for each specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: International Units/milliliter (IU/mL)
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 73 | 81 | 76 | 59 | 44 | 35
International Units/milliliter (IU/mL)
  At age of 5 months: number analyzed (Participants) | 0 | 0 | 76 | 0 | 0 | 0
  At age of 5 months |  |  | 0.9 [0.7 to 1.1] |  |  |
  At age of 7 months: number analyzed (Participants) | 73 | 81 | 0 | 59 | 44 | 35
  At age of 7 months | 1.7 [1.4 to 2.0] | 1.9 [1.6 to 2.2] |  | 1.6 [1.3 to 2.0] | 1.3 [1.1 to 1.7] | 1.5 [1.1 to 1.9]

32. Primary Outcome: Geometric Mean Concentrations of Antibodies to Tetanus Toxoid: Groups 1, 2, 3, 4, 6, and 7 - Booster Per-Protocol Population
Description: Antibody concentrations against tetanus toxoid were measured by ELISA and expressed as GMC. Booster PPP was defined as the PPP that was used for reporting data of time points at and after the age of 12 months. Here, '0' in number analyzed field signifies none of the participants were evaluable at that specified time point because different groups had different planned data collection time points as defined in time frame and pre-specified in protocol.
Time Frame: Groups 1, 3, 4, and 6: at the age of 13 months, Group 2 and 7: at the age of 16 months
Population: Analysis was performed on Booster PPP. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure and 'Number analyzed'=participants with available data for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 58 | 64 | 54 | 46 | 25 | 26
IU/mL
  At age of 13 months: number analyzed (Participants) | 58 | 0 | 54 | 46 | 25 | 0
  At age of 13 months | 1.8 [1.4 to 2.3] |  | 2.2 [1.8 to 2.8] | 1.7 [1.3 to 2.2] | 0.2 [0.2 to 0.4] |
  At age of 16 months: number analyzed (Participants) | 0 | 64 | 0 | 0 | 0 | 26
  At age of 16 months |  | 5.1 [4.1 to 6.3] |  |  |  | 2.7 [2.0 to 3.6]

33. Primary Outcome: Geometric Mean Concentrations of Antibodies to Tetanus Toxoid: Group 5 - Per-Protocol Population
Description: Antibody concentrations against tetanus toxoid were measured by ELISA and expressed as GMC.
Time Frame: At the age of 13 months
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 5: MenACYW Conjugate Vaccine: 12 Months
Number analyzed (Participants) | 56
IU/mL | 2.3 [1.8 to 3.1]

34. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: Solicited injection site reactions: tenderness/pain, erythema, and swelling and were planned to be collected and reported for each vaccine separately and not planned to be collected for Rotavirus vaccine. Here, '0' in number analyzed field for MenACYW categories signifies no participant were evaluable because in Groups 6 and 7 MenACYW vaccine was not administered; for Group 5, '0' in number analyzed field signifies safety data collection was not planned for Pentacel and Hepatitis-B vaccines; for Groups 2 and 7, '0' in number analyzed field signifies safety data collection was not planned for M-M-RII and VARIVAX vaccines, as pre-specified.
Time Frame: Within 7 days post any vaccination
Population: Analysis was performed on safety population that included participants who received at least 1 dose of investigation vaccine and for whom safety data were available. Here, 'Number analyzed'=participants with available data for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 5: MenACYW Conjugate Vaccine: 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 104 | 102 | 100 | 74 | 70 | 52 | 49
Participants
  MenACYW conjugate vaccine: Tenderness: number analyzed (Participants) | 100 | 99 | 100 | 73 | 68 | 0 | 0
  MenACYW conjugate vaccine: Tenderness | 76 | 78 | 70 | 49 | 29 |  |
  MenACYW conjugate vaccine: Erythema: number analyzed (Participants) | 100 | 99 | 100 | 73 | 68 | 0 | 0
  MenACYW conjugate vaccine: Erythema | 46 | 45 | 32 | 31 | 18 |  |
  MenACYW conjugate vaccine: Swelling: number analyzed (Participants) | 100 | 99 | 100 | 73 | 68 | 0 | 0
  MenACYW conjugate vaccine: Swelling | 29 | 28 | 21 | 21 | 11 |  |
  Pentacel: Tenderness: number analyzed (Participants) | 100 | 99 | 100 | 73 | 0 | 49 | 48
  Pentacel: Tenderness | 69 | 77 | 62 | 40 |  | 32 | 36
  Pentacel: Erythema: number analyzed (Participants) | 100 | 99 | 100 | 73 | 0 | 49 | 48
  Pentacel: Erythema | 41 | 45 | 21 | 20 |  | 21 | 25
  Pentacel: Swelling: number analyzed (Participants) | 100 | 99 | 100 | 73 | 0 | 49 | 48
  Pentacel: Swelling | 28 | 37 | 18 | 14 |  | 15 | 17
  Prevnar or Prevnar 13: Tenderness: number analyzed (Participants) | 100 | 99 | 100 | 73 | 68 | 49 | 48
  Prevnar or Prevnar 13: Tenderness | 74 | 69 | 72 | 51 | 32 | 36 | 38
  Prevnar or Prevnar 13: Erythema: number analyzed (Participants) | 100 | 99 | 100 | 73 | 68 | 49 | 48
  Prevnar or Prevnar 13: Erythema | 47 | 43 | 38 | 33 | 14 | 26 | 19
  Prevnar or Prevnar 13: Swelling: number analyzed (Participants) | 100 | 99 | 100 | 73 | 68 | 49 | 48
  Prevnar or Prevnar 13: Swelling | 35 | 33 | 25 | 28 | 12 | 21 | 15
  Hepatitis-B: Tenderness: number analyzed (Participants) | 99 | 98 | 92 | 73 | 0 | 48 | 47
  Hepatitis-B: Tenderness | 60 | 64 | 49 | 38 |  | 32 | 30
  Hepatitis-B: Erythema: number analyzed (Participants) | 99 | 98 | 92 | 73 | 0 | 48 | 47
  Hepatitis-B: Erythema | 34 | 22 | 14 | 17 |  | 21 | 13
  Hepatitis-B: Swelling: number analyzed (Participants) | 99 | 98 | 92 | 73 | 0 | 48 | 47
  Hepatitis-B: Swelling | 23 | 17 | 12 | 8 |  | 15 | 10
  M-M-RII: Tenderness: number analyzed (Participants) | 71 | 0 | 78 | 60 | 68 | 41 | 0
  M-M-RII: Tenderness | 29 |  | 39 | 26 | 31 | 25 |
  M-M-RII: Erythema: number analyzed (Participants) | 71 | 0 | 78 | 60 | 68 | 41 | 0
  M-M-RII: Erythema | 16 |  | 16 | 14 | 8 | 12 |
  M-M-RII: Swelling: number analyzed (Participants) | 71 | 0 | 78 | 60 | 68 | 41 | 0
  M-M-RII: Swelling | 10 |  | 11 | 9 | 7 | 6 |
  VARIVAX: Tenderness: number analyzed (Participants) | 71 | 0 | 78 | 60 | 68 | 41 | 0
  VARIVAX: Tenderness | 27 |  | 36 | 26 | 29 | 27 |
  VARIVAX: Erythema: number analyzed (Participants) | 71 | 0 | 78 | 60 | 68 | 41 | 0
  VARIVAX: Erythema | 17 |  | 13 | 17 | 12 | 14 |
  VARIVAX: Swelling: number analyzed (Participants) | 71 | 0 | 78 | 60 | 68 | 41 | 0
  VARIVAX: Swelling | 6 |  | 9 | 7 | 6 | 7 |

35. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: An solicited reaction (SR) was an adverse reaction (AR) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the electronic case report form (eCRF). Systemic AEs were all AEs that were not injection site reactions. They, therefore, include systemic manifestations as well as localized or topical manifestations that were not associated with the vaccination site. Solicited systemic reactions included Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability.
Time Frame: Within 7 days post any vaccination
Population: Analysis was done on safety population. Here, 'Number analyzed'=participants with available data for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 5: MenACYW Conjugate Vaccine: 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 104 | 102 | 100 | 74 | 70 | 52 | 49
Participants
  Fever: number analyzed (Participants) | 99 | 100 | 100 | 72 | 68 | 50 | 48
  Fever | 32 | 42 | 42 | 28 | 11 | 19 | 22
  Vomiting: number analyzed (Participants) | 101 | 100 | 100 | 73 | 68 | 49 | 48
  Vomiting | 28 | 33 | 27 | 10 | 8 | 14 | 12
  Crying abnormal: number analyzed (Participants) | 101 | 100 | 100 | 73 | 68 | 49 | 48
  Crying abnormal | 78 | 74 | 77 | 45 | 30 | 37 | 35
  Drowsiness: number analyzed (Participants) | 101 | 100 | 100 | 73 | 68 | 49 | 48
  Drowsiness | 71 | 81 | 75 | 46 | 30 | 37 | 38
  Appetite lost: number analyzed (Participants) | 101 | 100 | 100 | 73 | 68 | 49 | 48
  Appetite lost | 55 | 65 | 49 | 36 | 22 | 27 | 27
  Irritability: number analyzed (Participants) | 101 | 100 | 100 | 73 | 68 | 49 | 48
  Irritability | 86 | 92 | 88 | 63 | 48 | 44 | 42

36. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE was an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or onset post-vaccination. These included both serious and non-serious events.
Time Frame: Within 30 days post any vaccination
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 5: MenACYW Conjugate Vaccine: 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 104 | 102 | 100 | 74 | 70 | 52 | 49
Participants | 83 | 81 | 72 | 50 | 35 | 44 | 38

37. Primary Outcome: Number of Participants With Immediate Unsolicited AE
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE was an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or onset post-vaccination. These included both serious and non-serious events. Immediate Unsolicited AE were AEs reported within 30 minutes of vaccine administration.
Time Frame: Within 30 minutes post any vaccination
Population: Analysis was done on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 5: MenACYW Conjugate Vaccine: 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
Number analyzed (Participants) | 104 | 102 | 100 | 74 | 70 | 52 | 49
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited non-serious AEs were collected from Day 0 to Day 30 post any vaccination. SRs were collected within 7 days post any vaccination. Serious adverse events were collected throughout the trial (up to the age of 13 months for Groups 1, 3, 4, 5 and 6; up to the age of 16 months for Groups 2 and 7), i.e. 30 days after last vaccination.
Description: SR: an AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was done on safety population. In the AE section, solicited reactions Fever, Crying abnormal, Drowsiness, and Appetite lost are reported under Pyrexia, Crying, Somnolence, and Anorexia, respectively.
Arm/Group | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months | Group 5: MenACYW Conjugate Vaccine: 12 Months | Group 6: Control: 2, 4, 6, and 12 Months | Group 7: Control: 2, 4, 6, 12, and 15 Months
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/102 | 0/100 | 2/74 | 0/70 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/104 | 5/102 | 7/100 | 5/74 | 1/70 | 4/52 | 4/49
Other Adverse Events (participants affected / at risk) | 99/104 | 98/102 | 98/100 | 71/74 | 59/70 | 51/52 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months (N=104) | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months (N=102) | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months (N=100) | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months (N=74) | Group 5: MenACYW Conjugate Vaccine: 12 Months (N=70) | Group 6: Control: 2, 4, 6, and 12 Months (N=52) | Group 7: Control: 2, 4, 6, 12, and 15 Months (N=49)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kawasaki's Disease (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine: 2, 4, 6, and 12 Months (N=104) | Group 2: MenACYW Conjugate Vaccine: 2, 4, 6, and 15 Months (N=102) | Group 3: MenACYW Conjugate Vaccine: 2, 4, and 12 Months (N=100) | Group 4: MenACYW Conjugate Vaccine: 6 and 12 Months (N=74) | Group 5: MenACYW Conjugate Vaccine: 12 Months (N=70) | Group 6: Control: 2, 4, 6, and 12 Months (N=52) | Group 7: Control: 2, 4, 6, 12, and 15 Months (N=49)
Conjunctivitis (Eye disorders) | 4 (4) | 8 (8) | 0 (0) | 5 (5) | 2 (2) | 3 (3) | 7 (7)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3) | 5 (5) | 2 (2) | 0 (0) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 8 (9) | 5 (7) | 6 (6) | 4 (4) | 2 (2) | 4 (5)
Flatulence (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (5) | 3 (3) | 0 (0) | 5 (7) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 (5) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Teething (Gastrointestinal disorders) | 13 (27) | 10 (16) | 7 (9) | 7 (17) | 2 (2) | 5 (13) | 4 (10)
Vomiting (Gastrointestinal disorders) | 29 (42) | 35 (46) | 28 (46) | 11 (14) | 8 (8) | 14 (19) | 16 (19) — Vomiting events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Injection Site Erythema (General disorders) | 59 (324) | 57 (269) | 48 (188) | 44 (153) | 24 (54) | 30 (153) | 27 (92)
Injection Site Haematoma (General disorders) | 11 (23) | 5 (5) | 6 (13) | 8 (10) | 1 (1) | 3 (5) | 3 (3)
Injection Site Pain (General disorders) | 82 (594) | 83 (626) | 79 (509) | 57 (272) | 40 (121) | 37 (297) | 39 (219)
Injection Site Swelling (General disorders) | 46 (185) | 45 (165) | 32 (135) | 39 (95) | 17 (38) | 24 (90) | 21 (71)
Irritability (General disorders) | 86 (223) | 92 (251) | 88 (189) | 63 (100) | 48 (48) | 44 (126) | 42 (116)
Pyrexia (General disorders) | 38 (61) | 46 (79) | 46 (66) | 31 (34) | 14 (15) | 21 (32) | 22 (42) — Pyrexia/Fever events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Bronchiolitis (Infections and infestations) | 5 (7) | 5 (7) | 6 (7) | 5 (5) | 2 (2) | 4 (5) | 0 (0)
Candidiasis (Infections and infestations) | 4 (5) | 6 (6) | 6 (6) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Croup Infectious (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 5 (5)
Otitis Media (Infections and infestations) | 29 (43) | 21 (31) | 20 (23) | 20 (24) | 8 (9) | 13 (18) | 21 (25)
Otitis Media Acute (Infections and infestations) | 6 (7) | 12 (22) | 4 (4) | 4 (6) | 1 (1) | 3 (3) | 2 (3)
Sinusitis (Infections and infestations) | 6 (6) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 31 (40) | 36 (46) | 15 (16) | 15 (19) | 3 (3) | 18 (23) | 18 (20)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 55 (93) | 65 (107) | 49 (75) | 36 (45) | 22 (22) | 27 (54) | 27 (43)
Crying (Nervous system disorders) | 78 (164) | 74 (173) | 77 (137) | 45 (66) | 30 (30) | 38 (93) | 35 (77) — Crying/Crying abnormal events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Somnolence (Nervous system disorders) | 71 (142) | 81 (176) | 75 (137) | 46 (60) | 30 (30) | 37 (87) | 38 (77)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 13 (15) | 6 (6) | 3 (4) | 2 (2) | 3 (5) | 7 (7)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (9) | 6 (8) | 0 (0) | 1 (1) | 6 (6) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (9) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 2 (2)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 3 (4)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.